CLINICAL TRIAL: NCT00918762
Title: A Pilot Study Assessing the Use of DA VINCI® Robotic Surgical System in Laryngeal and Pharyngeal Surgeries
Brief Title: Transoral Robotic Surgery or Standard Surgery in Treating Patients With Benign or Malignant Tumors of the Larynx and Pharynx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ho-Sheng Lin, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000642940; P30CA022453 (NIH); WSU-2008-022
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Head and Neck Cancer; Perioperative/Postoperative Complications; Precancerous Condition
Keywords: perioperative/postoperative complications; precancerous condition; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Postoperative Complications; Precancerous Conditions; Squamous Cell Carcinoma of Head and Neck | interventions — Video-Assisted Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- daVinci® Robotic Surgical System (Experimental): Participants will undergo a planned surgical procedures via the robotic approach.
  Interventions: Procedure: assessment of therapy complications; Procedure: diagnostic endoscopic surgery; Procedure: quality-of-life assessment; Procedure: therapeutic conventional surgery; Procedure: therapeutic endoscopic surgery; Procedure: transoral robotic surgery; Procedure: video-assisted surgery

INTERVENTIONS:
Procedure: assessment of therapy complications
Procedure: diagnostic endoscopic surgery
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery
Procedure: therapeutic endoscopic surgery
Procedure: transoral robotic surgery
Procedure: video-assisted surgery

SUMMARY:
RATIONALE: Transoral robotic surgery may make it easier to find and remove benign or malignant tumors of the larynx and pharynx and cause less damage to normal tissue. It is not yet known whether transoral robotic surgery is more effective than standard surgery in diagnosing and treating larynx and pharynx tumors.

PURPOSE: This phase I trial is studying how well transoral robotic surgery works compared with standard surgery in treating patients with benign or malignant tumors of the larynx or pharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the potential benefits of using the transoral robotic surgical approach against the conventional open and transoral approaches in patients with benign or malignant disease involving the larynx and pharynx.

Secondary

* Determine the proportion of laryngeal and pharyngeal surgical procedures where the surgical exposure is adequate to allow the successful completion of the surgical resection using the transoral robotic surgical approach.

OUTLINE: Patients are assigned to transoral robotic surgery or standard therapy consisting of conventional transoral endoscopic or open approach according to their preference.

Patients undergo planned surgical procedures (either diagnostic or therapeutic) appropriate for their disease in the larynx or pharynx via the transoral robotic surgical approach or the conventional transoral endoscopic or open approach.

Patients complete the Functional Assessment of Cancer Therapy Head and Neck Scale, the Performance Status Scale for Head and Neck Cancer Patients, and the University of Washington Quality of Life Scale at baseline and at 3 and 6 months. Patients also undergo voice analysis by acoustic analyses, and speech and swallow pathology evaluation by videostroboscopy and modified barium swallow.

After completion of study procedure, patients are followed at 3 and 6 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued to the control group (standard conventional surgery) and 30 patients will be accrued to the robotic surgery group.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Benign or malignant disease of the larynx or pharynx that requires surgical intervention for either diagnostic or therapeutic purposes

  * Malignant disease must meet the following criteria:

    * Histologically confirmed diagnosis of 1 of the following:

      * Glottic cancer (T1, T2, and T3)
      * Supraglottic cancer (T1, T2, and T3)
      * Hypopharyngeal cancer (T1 and T2)
      * Oropharyngeal cancer (T1, T2, and T3)
      * Nasopharyngeal cancer (T1 and T2)
    * Resectable involved lymph nodes
    * No invasion of osseous and/or osseocartilaginous structures including the following:

      * Mandibular bone
      * Thyroid cartilage
      * Hyoid bone
      * Cricoid bone
      * Vertebral body
    * No pharyngeal wall or tongue-based involvement requiring resection of > 50% of the posterior pharyngeal wall or tongue base
    * No radiological confirmation of carotid artery involvement
    * No fixation of tumor to the prevertebral fascia
    * No bilateral arytenoid involvement
    * No surgical defect requiring open approach for reconstruction
    * No evidence of distant metastasis

PATIENT CHARACTERISTICS:

* Not pregnant
* No unexplained fever and/or untreated active infection
* No medical conditions contraindicating general anesthesia
* No inadequate jaw opening due to prior head and neck surgery, trauma, or radiotherapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Operative time that directly affects operative cost | post operative

SECONDARY OUTCOMES:
Blood loss | During surgery
Intra-operative and post-operative complications | during the operation and post operative
Need for reconstruction | post operative
Margins status | post operative
Length of hospital stay | during time as inpatient
Tracheostomy and PEG dependence | post operative
Days to oral intake | post operative
Time to locoregional recurrence | post operative
Speech intelligibility | post operative
Quality of life | 3 months and 6 month following completion of surgery
Postoperative pain | post operative
Proportion of robotic surgical cases where adequate surgical exposure allowed for successful operation completion | post operative

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Sheng Lin, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States